CLINICAL TRIAL: NCT07378735
Title: Back to Life - Early Rehabilitation Therapy for Patients Undergoing Lumbar Spinal Fusion Surgery - A Single-case Experimental Design Study
Brief Title: Back to Life - Early Rehabilitation Therapy for Patients Undergoing Lumbar Spinal Fusion - A Single-case Experimental Study
Acronym: Back to Life
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Health Care Centre Frederiksberg (Unknown); The Danish Arthritis Association (Unknown); The Capital Region of Denmark Research Foundation (Unknown); Lundbeck Foundation (Other); Danish Physiotherapists (Unknown); The Cross-Sectoral Fund (Unknown)
Responsible Party: Principal Investigator, Heidi Tegner, Research Physiotherapist, Post doc, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-25053000; p-2024-17807 (Other: The Danish Data Protection Agency)
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Low Back Pain; Lumbar Spinal Fusion
Keywords: Physical activity; Low back pain; Lumbar spinal fusion; Exercise; Rehabilitation; Physiotherapy; Single-case experimental study; Cognitive behavioural approach
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Intervention Model Description: The study is a single-case experimental study using a Multiple Baseline Design. A characteristic of Multiple Baseline Design is the manipulation of the intervention by introducing it at different points in time. Therefore, the cognitive-behavioural approach will start at 14, 18, 22, and 26 days post-surgery, respectively.
Who Masked: Investigator
Masking Description: Full blinding is not feasible in this MBD. Allocation to baseline length will be concealed until the intervention is initiated. The randomisation schedule will be generated by co-investigator Jan Christensen.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SOGA - 14 days post-surgery (Active Comparator): The intervention SOGA will start 14 days after the participants lumbar spinal fusion.
  Interventions: Behavioral: SOGA - Socratic dialogue and Graded Activity
- SOGA - 18 days post-surgery (Active Comparator): The intervention SOGA will start 18 days after the participants lumbar spinal fusion.
  Interventions: Behavioral: SOGA - SOcratic dialougue and Graded-Activity
- SOGA - 22 days post-surgery (Active Comparator): The intervention SOGA will start 22 days after the participants lumbar spinal fusion.
  Interventions: Behavioral: SOGA - SOcratic dialogue and Graded-Activity
- SOGA - 26 days post-surgery (Active Comparator): The intervention SOGA will start 28 days after the participants lumbar spinal fusion.
  Interventions: Behavioral: SOGA - SOcratic dialogue and Graded Activity

INTERVENTIONS:
Behavioral: SOGA - Socratic dialogue and Graded Activity — SOGA consists of six sessions over two months and is based on a cognitive behavioural approach, starting 14 days after surgery. The intervention is delivered through home visits, in-person sessions at Frederiksberg Health Care Centre, and telephone consultations.
  The content includes dialogue and exercise, specifically SOcratic dialogue and Graded Activity (in short called SOGA). The dialogue alternates between a deductive approach based on knowledge exchange between the physiotherapist and the participant and an inductive approach using Socratic dialogue. Socratic dialogue involves guided questioning, summaries, and reflections to support the participant's understanding of pain, surgery, and physical activity and to encourage the participant to form their own conclusions. Graded activity is based on operant conditioning principles and uses structured exercise progression to increase meaningful activity levels and reduce pain-related behaviours despite the presence of pain.
  Arms: SOGA - 14 days post-surgery
Behavioral: SOGA - SOcratic dialougue and Graded-Activity — SOGA consists of six sessions over two months and is based on a cognitive behavioural approach, starting 18 days after surgery. The intervention is delivered through home visits, in-person sessions at Frederiksberg Health Care Centre, and telephone consultations.
  The content includes dialogue and exercise, specifically SOcratic dialogue and Graded Activity (in short called SOGA). The dialogue alternates between a deductive approach based on knowledge exchange between the physiotherapist and the participant and an inductive approach using Socratic dialogue. Socratic dialogue involves guided questioning, summaries, and reflections to support the participant's understanding of pain, surgery, and physical activity and to encourage the participant to form their own conclusions. Graded activity is based on operant conditioning principles and uses structured exercise progression to increase meaningful activity levels and reduce pain-related behaviours despite the presence of pain.
  Arms: SOGA - 18 days post-surgery
Behavioral: SOGA - SOcratic dialogue and Graded-Activity — SOGA consists of six sessions over two months and is based on a cognitive behavioural approach, starting 22 days after surgery. The intervention is delivered through home visits, in-person sessions at Frederiksberg Health Care Centre, and telephone consultations.
  The content includes dialogue and exercise, specifically SOcratic dialogue and Graded Activity (in short called SOGA). The dialogue alternates between a deductive approach based on knowledge exchange between the physiotherapist and the participant and an inductive approach using Socratic dialogue. Socratic dialogue involves guided questioning, summaries, and reflections to support the participant's understanding of pain, surgery, and physical activity and to encourage the participant to form their own conclusions. Graded activity is based on operant conditioning principles and uses structured exercise progression to increase meaningful activity levels and reduce pain-related behaviours despite the presence of pain.
  Arms: SOGA - 22 days post-surgery
Behavioral: SOGA - SOcratic dialogue and Graded Activity — SOGA consists of six sessions over two months and is based on a cognitive behavioural approach, starting 26 days after surgery. The intervention is delivered through home visits, in-person sessions at Frederiksberg Health Care Centre, and telephone consultations.
  The content includes dialogue and exercise, specifically SOcratic dialogue and Graded Activity (in short called SOGA). The dialogue alternates between a deductive approach based on knowledge exchange between the physiotherapist and the participant and an inductive approach using Socratic dialogue. Socratic dialogue involves guided questioning, summaries, and reflections to support the participant's understanding of pain, surgery, and physical activity and to encourage the participant to form their own conclusions. Graded activity is based on operant conditioning principles and uses structured exercise progression to increase meaningful activity levels and reduce pain-related behaviours despite the presence of pain.
  Arms: SOGA - 26 days post-surgery

SUMMARY:
Aim This study aims to assess the effectiveness of an early intervention comprising individually tailored physiotherapy, including dialogue, education, and graded activity, following lumbar spinal fusion surgery. The effectiveness will be evaluated on patient-specific goals, physical activity, pain intensity, pain interference, fear of movement, and pain self-efficacy for patients after a lumbar spinal fusion.

DETAILED DESCRIPTION:
In 2023, above 1400 patients underwent lumbar spinal fusion (LSF) in Denmark to treat CLBP. LSF aims to relieve pain by eliminating movement between joints by fusing one or more adjacent vertebrae. The use of LSF has been increasing because of the ageing population and because of improvements in surgical techniques and technologies.

Unfortunately, despite LSF surgery, many patients are not improving their physical activity level post-surgery, and inactivity is associated with an increased risk of disease mortality.

Therefore, healthcare professionals must address physical activity in post-surgical rehabilitation to help patients achieve healthy behaviour after surgery.

To perform physical activity, both physiological, psychological, and social factors have an influence. Further, qualitative interviews with patients undergoing LSF reveal significant concerns about engaging in physical activity after surgery. It thereby seems important that a rehabilitation approach includes a bio-psycho-social approach to incorporate the complexity of physical activity.

Rehabilitation involving physical exercises combined with a cognitive behavioural approach (CBA) has shown beneficial effects on short- and long-term functional outcomes in patients undergoing LSF. The purpose of CBA is to provide patients with techniques that can lead to a sense of control over their lives, despite pain. The approaches have no sharply defined treatment modalities but include a range of techniques that modify the behavioural, cognitive, affective, and sensory aspects of pain. Tegner et al. supported the evidence of a CBA in an RCT by showing that CBA was safe to start with just after LSF and significantly affected fear of movement and sedentary behaviour compared to usual care.

Despite the increasing consensus regarding an early CBA for patients after LSF, several problems remain unsolved. First, in many studies, the beneficial effect of an early approach consisting of CBA post-surgery is not above the minimal clinically important change.

Secondly, a huge concern is that rehabilitation, including CBA, is complex and time-consuming and thereby difficult to implement in a clinical setting where time and resources are sparse. Thirdly, it is still uncertain what drives the beneficial effects of CBA, what constitutes optimal intervention timing, and which components moderate and mediate change in physical activity behaviour.

To investigate these problems, several initiatives are needed, among others, the use of alternative research methods which include the individual patients much closer. Furthermore, a close collaboration between health sectors is important to integrate each responsible partner in the rehabilitation process, to incorporate the essential expertise and experience, and finally to be able to design an intervention that is realistic and manageable to implement in clinical practice.

Therefore, in this project, the investigators will implement an early CBA in close collaboration between partners from the hospital and a rehabilitation centre. Further, the investigators would like to test the effect of the intervention closely on patients after surgery based on function, physical activity and pain response by a single-case experimental study design (SCED) in the setting where the rehabilitation in clinical practice will be performed.

Aim and hypothesis This study aims to test the effectiveness of an early intervention consisting of a CBA on a patient-specific goal, physical activity, pain intensity, pain interference, fear of movement, and pain self-efficacy for patients after an LSF. An intervention planned between sectors and delivered in a community care centre.

ELIGIBILITY:
The investigators will in total include 12 patients undergoing an LSF from the Centre for Rheumatology and Spine Diseases at Rigshospitalet, Denmark.

Before inclusion, a pilot of three participants will be performed.

Inclusion Criteria for all included:

* ≥ 18 years of age
* Low back pain (LBP) > 3 months
* Read and understand the Danish language
* The participants should be a part of Frederiksberg Municipality and Copenhagen Municipality (in Denmark)

Exclusion Criteria:

* Post-traumatic vertebral compression/deformity
* Patients with the following conditions (infection, neoplasm, metastasis, metabolic bone disease, fractures or other known autoimmune arthropathies)
* Patients with patient-related circumstances (physical or mental status) that impede their ability to give informed consent and adhere to the study program (e.g., dementia, developmental disorders, or substance-induced cognitive impairment)
* Other special conditions, where the patient is judged by the surgeon as inappropriate to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Patient-specific goal | Daily, from 1 day post-surgery to 3 months post-surgery
  The patient-specific goal will be reported as the primary outcome. To evaluate the participants' ability to reach their overall goal of the surgery and following rehabilitation, the participants are asked, together with the PI, to formulate an individualised, measurable, achievable, realistic/relevant, and time-bound (SMART) goal. The goal should be manageable to achieve within the three-month intervention period. The participant will evaluate their ability to reach their goal on a scale from 0 ('unable to do') to 10 ('able to perform at the same level as before the injury or problem).

SECONDARY OUTCOMES:
Physical activity | Daily, from 1 day post-surgery to 3 months post-surgery
  Physical activity is defined as any bodily movement produced by skeletal muscles that requires energy expenditure. Physical activity thereby refers to all movement, including low-, moderate- and vigorous-intensity physical activity. Total physical activity will be the main physical activity outcome; however, steps per day and light, moderate, and vigorous physical activity will be reported for exploratory purposes.
  To measure the amount of time doing physical activity per day, we will use activity data from the accelerometers from the SENS Motion activity measurement system. The accelerometer will be fastened on the thigh using a band-aid that does not interfere with everyday activities. Data will be collected via a dedicated smartphone application installed on the participant's smartphone that automatically uploads data to a secure server but does not provide any data to the participant.
Pain intensity | Daily, from 1 day post-surgery to 3 months post-surgery
  Patient-reported LBP intensity will in this study be defined as "The present pain in the area on the posterior aspect of the body from the lower margin of the twelfth ribs to the lower gluteal folds with or without pain referred into one or both lower limbs".
  LBP intensity will be measured by the 11-point numerical rating scale (NRS), rating from 0 representing no pain to 10 representing the worst pain imaginable pain
Fear of movement | Daily, from 1 day post-surgery to 3 months post-surgery
  Fear of movement will be measured by the physical activity component of the Fear-Avoidance Beliefs Questionnaire (FABQ-P). FABQ-P includes five statements answered by a score from strongly disagree (0 on a Likert scale) to strongly agree (6 on a Likert scale). The FABQ has acceptable internal consistency, test-retest reliability, and construct validity. Further, the responsiveness of the FABQ-PA is moderate in an acute LBP sample. The FABQ has been translated into Danish.
Pain interference | Daily, from 1 day post-surgery to 3 months post-surgery
  Pain interference is defined as the consequences of pain on relevant aspects of a patient's life. This includes the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities. Further pain interference also includes problems with sleep and enjoyment of life. For this study, pain interference will be based on two variables by asking the participants to rate daily, on a scale ranging from 0 ("Has not affected at all") to 10 ("Has affected to the greatest extent"), to what extent pain has interfered with their "movement in daily life" and "enjoyment of life" The two aspects of pain interference have been chosen among the above broad definition of pain interference based on a validated survey among 30 patients going through LSF assessed by the principal investigator and colleagues.
Pain self-efficacy | Daily, from 1 day post-surgery to 3 months post-surgery
  Self-efficacy is defined as a person's confidence or belief in the capacity to achieve goals and specific tasks. Pain self-efficacy is based on the definition of self-efficacy and reflects the patient's believed confidence in their ability to achieve specific goals and everyday activities, despite their pain. Patient-reported pain self-efficacy is measured using the short form of the Pain Self-efficacy Questionnaire (PSEQ-2). PSEQ-2 will be measured by the 7-point rating scale, ranging from 0 "Not at all confident" to 6 "Completely confident".

OTHER OUTCOMES:
Additional questions | Daily, from 1 day post-surgery to 3 months post-surgery
  Two additional questions will be asked each day, including a free-text area:
  1. Have you taken more or less pain medication, and if yes, please briefly explain why?
  2. Has anything happened in the past 24 hours, apart from your normal daily routine, that has affected your physical activity or pain? If yes, please briefly explain what has affected your physical activity or pain.

CONTACTS AND LOCATIONS:
Overall Officials: Bente Appel Esbensen, Professor, Study Chair — Centre for Rheumatology and Spine Diseases, Rigshospitalet

IPD SHARING:
Plan to Share IPD: Yes
On reasonable request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting 6 months after publication
Access Criteria: De-identified individual participant data will be shared with qualified researchers who have a scientifically relevant research question. Data sharing will be subject to approval of a written research proposal describing the planned analyses. Access will require the signing of a data sharing agreement outlining the purpose of use, data protection, and confidentiality. Requests can be submitted by contacting the study investigators.